CLINICAL TRIAL: NCT02496299
Title: Comparison Of The Effect Of Dexamethasone Added To Bupivacaine With Plain Bupivacaine For Caudal Block In Patients For Herniotomy.
Brief Title: Effect of Dexamethasone Added To Bupivacaine During Caudal Block
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lagos State University (Other)
Responsible Party: Principal Investigator, FAGBOHUN ADUNNI OMOLOLA, Dr, Lagos State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SAS 022015
Record Dates: First submitted 2015-07-05; First posted 2015-07-14 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Caudal Block
Keywords: COMPARISSON; CAUDAL BLOCK; BUPIVACAINE; DEXAMETHASONE
MeSH Terms: interventions — Dexamethasone; Steroids; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexametasone (BD), (Active Comparator): BD ,a mixture of 0.2mg/kg dexamethasone in 1ml/kg bupivacaine
  Interventions: Drug: Dexamethasone
- Bupivacaine,B (Active Comparator): B ,1ml/kg bupivacaine:
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone — Comparison of analgesic effects of dexamethasone with plain bupivacaine during caudal blocks in children
  Other Names: STEROID,LOCAL ANAEDSTHETIC
  Arms: dexametasone (BD),
Drug: Bupivacaine — Comparison of analgesic effects of dexamethasone with plain bupivacaine during caudal blocks in children
  Other Names: heavy marcaine
  Arms: Bupivacaine,B

SUMMARY:
It is a prospective double blind randomized study on the effect of dexamethasone added to bupivacaine with plain bupivacaine for caudal block in patient for herniotomy.

96 patients between the ages 1-6 years will be randomly selected and divided into two groups; B and BD.

Group B will receive 1ml/kg bupivacaine 0.25% (maximum volume 20mls) and group BD will receive a mixture of 0.2mg/kg dexamethasone in 1ml/kg bupivacaine 0.25% (maximum volume = 20mls).

Data taken will then be analyzed and interpreted.

DETAILED DESCRIPTION:
METHODOLOGY STUDY DESIGN. The study will be a prospective study. All the patients will be randomized into two groups, B and BD. In group B, patients will receive 1 ml/kg bupivacaine 0.25% (maximum volume = 20 ml). In group BD, patients will receive a mixture of 0.2 mg/kg dexamethasone in 1 ml/kg bupivacaine 0.25% (maximum volume = 20 ml). The total volume injected will be 1 ml/kg in all patients.

RESEARCH SETTING. The study will take place at Gbagada, Alimosho and Ifako Ijaye General Hospitals in Lagos.

They are all secondary health care facilities with 800 bed spaces in Gbagada, 400 at Alimosho and 300 at Ifako Ijaye. General Hospital Gbagada was established in 1983 and situated in Gbagada, Alimosho in 2006, situated at Igando while Ifako ijaye was created in 2005 and located at Ifako. These three areas are densely populated suburbs of Lagos.

SAMPLE SIZE ESTIMATION. The minimum sample size for this study was calculated with the formula below 21

n= z 2 x p x q d2 Assuming a 95% interval, 5% level of precision and a proportion of 90% 21 .

Where n =minimum sample size Z =a constant (1.96 ;) a percentage point on standard normal deviation corresponding to 95% confidence interval.

P =proportion of patient with positive dexamethasone analgesic effect obtained from a past study. (90%) 21 Q = complimentary probability; equivalent to (1-p) d =predetermined level of precision equivalent to 5% n= (1.96) 2 x 0.90 x.055 0.05 =76.0 approximated to 80 Sample size will be increased by 20% to provide for attrition=16 Therefore, sample size will be 80+16=96

RANDOMIZATION After local ethics committee approval and a written informed consent has been obtained from parents or legal guardians, 96 patients undergoing elective unilateral inguinal herniotomy will be selected for this prospective randomized-controlled trial.

Patients would be distributed into two equal groups: group B (n = 48), in which the caudal block will be performed using only bupivacaine, and group BD (n = 48), in which the caudal block will be performed using dexamethasone added to bupivacaine. The distribution will be by simple randomization method using computer generated random numbers.

Numbers 1-96 will be randomly distributed into the two groups with each group having a total of 48 patients.

ALLOCATION CONCEALMENT MECHANISM The patients will be seen at least a day before surgery for preoperative assessment.

All patients would be fasted according to the AMERICAN SOCIETY OF ANESTHESIOLOGY (ASA) guidelines (2 h for clear fluids; 4 h for breast milk; 6 h for formula milk or light meal). No premedication will be administered and an informed written consent form will be filled by parent or guardian after adequate explanation of the scope of the study to parent or guardian and the older child as the case may be.

All patients will have routine investigations performed. There will be two residents recruited as research assistants.Post emergence, the first ,assistant(who is also unaware of the group allocation)is to observe patient in the recovery room post operatively hence methods of pain assessment post operatively will be discussed with this research assistant.

The second research assistant assigns participants to interventions and prepares the drugs. This assistant stays outside the operating room but within the theatre environ as he holds the key to the code.

Using the sealed envelope technique, numbers 1-96 is placed in an envelope from which a research assistant allows patients parent or legal guardian to randomly pick a number.

The research assistant then compares with the computer generated random sequence to determine which of the groups the patient belongs.

Both the patient and investigator will be blinded to the allocation. All drugs will be prepared aseptically by this research assistant. The assistant would prepare the drugs. On arrival at the operating room, routine standard monitors would be applied (Electrocardiograph, noninvasive blood pressure, and pulse oximetry) and baseline vital signs taken.

General anesthesia would be induced by the investigator (who is unaware of the group allocation) with incremental dose of halothane from 0.5- 2% in 100% oxygen. After induction of anesthesia, an intravenous line would be placed, followed by the insertion of an appropriately sized laryngeal mask airway which will be secured with tapes.

When an adequate depth of anesthesia is attained, anesthesia would be maintained using isoflurane 1-2% in 100% oxygen. No muscle relaxants will be administered and the patients would breathe spontaneously using Mapleson F till the end of surgery. After properly securing the laryngeal mask airway, patients will be turned to the left lateral position.

Under complete aseptic conditions caudal block will be performed using a 25-G short beveled needle. Correct placement of the needle will be confirmed by the characteristic 'pop' felt as the sacrococcygeal membrane when penetrated.

The stilet will be removed while the plastic cannula is secured. Correct placement in the epidural space will be confirmed by absence of cerebrospinal fluid flow and absence of swelling during injection of drugs which occurs with a subcutaneous insertion.

The investigator, who is the anesthesiologist performing the block would be blinded to the identity of the drug used as the epidural injectate for all patients would be presented in a 20 mls syringe containing 20mls of a colourless, odourless, non-particulate solution of which the investigator who is the performer of the caudal block gives a dose of 1ml/kg.

The codes B and BD are only known to the research assistant who prepared the drugs and only discloses the codes at the end of the study or in the event of an adverse reaction to any of the drugs used in the study.

The end of injection will be taken as zero time. Surgery would commence 10 min after the block is performed to allow for the drugs to take effect.

A standardized intraoperative fluid therapy will be used in all patients (10 ml/kg/h of normal saline solution). Mean arterial blood pressure (MAP), heart rate (HR), and arterial oxygen saturation (SpO2) would be recorded using non invasive blood pressure monitor and pulse oxymetry before induction and then every 5 min after induction of anesthesia till the end of surgery.

During the intraoperative period, adequacy of analgesia would be assessed by hemodynamic stability, which would be defined by the absence of an increase of more than 20% in HR or MAP compared with pre incision values. An increase of more than 20% in HR or MAP would be considered an indication of inadequate analgesia and managed by a bolus dose of intravenous paracetamol 15 mg/kg, followed by further doses of intravenous diclofenac 1mg/kg if needed. The need for intraoperative analgesics would be recorded.Such patient will be considered as part of attrition.

At the end of surgery, isoflurane is switched off and LMA is extubated when patient is awake.

Emergence time (the time from end of surgery to opening of the eyes on calling the patients name) and a delayed anesthetic emergence (considered if 20 minutes elapsed from the end of surgery to exiting the operating theatre) were noted.

After recovery, when the patients are able to maintain a patent airway, they would be transferred to the recovery room, where they remain for at least 2 h before being transferred to the ward. Post operative pain and hemodynamic variables (MAP and HR) would be recorded at the recovery room and then every 30 min till the patient is discharged to the ward after 3 hours. Postoperative pain will be assessed using a modified Objective Pain Score (mOPS) every 30 min for the first 2 h and at 4, 6, 8, 10, 12, 18, and 24 h postoperatively. This score includes five criteria: crying, agitation, movement, posture, and localization of pain. Each criterion is assigned a score from 0 to 2, with 2 being the worst, to yield a possible total score of 0-10 [5]. If the mOPS score is 4 or more, rescue analgesia in the form of paracetamol 15 mg/kg orally would be administered. Further boluses of paracetamol 15 mg/kg would be administered orally every 4 h if required.

Residual motor block and sedation level will be also assessed at 30 min and at 1, 2, 4, and 6 h after surgery. Motor block will be assessed using a modified Bromage scale consisting of four points [0 = full motor strength (flexion of knees and feet), 1 = flexion of knees, 2 = little movement of feet only, 3 = no movement of knees or feet] [29]. The sedation score will; be assessed using a four-point scale (1, alert and aware; 2, asleep, arousable by verbal contact; 3, asleep, arousable by physical contact; and 4, asleep, not arousable).

After transferring to the ward, rescue analgesia consumption, pain scores,the occurrence of postoperative vomiting during the first 24h after surgery will be recorded. Any other complications including itching, urine retention (no voiding of urine for 6 hour postoperative), respiratory depression (respiratory rate<10 breaths/min), hypotension (MAP decreased>20% of baseline), or bradycardia (HR decreased>20% of baseline) would be recorded by a research assistant for 24 hours. Any undesirable effect will be treated as follows; for shivering, patient is covered, given warm intravenous fluids, theatre room temperature is increased, for itching; intravenous chlorpheniramine is given, metoclopramide for vomiting, for urinary retention a catheter is passed.

The time to first supplemental oral paracetamol from the end of surgery to the first modified objective pain score of greater than or equal to 4 will be recorded.

The time to first micturition post caudal block and the incidence of bladder catheterization would also be recorded.

The postoperative data in the recovery room would be recorded by the second research assistant mentioned above, this is the second research assistant mentioned above, a resident who was also blinded to the drugs used during the caudal block.

The assistant would be with the patient in the recovery room for at least 3 hours before being transferred to the ward.

MEASUREMENT Data will be collected using a data collection form designed by the investigator.

Patients' blood pressure is measured with a noninvasive blood pressure monitor, heart rate and arterial oxygen saturation (SPO2) will be measured with a pulse oximeter and respiratory rate will be counted. These vital signs will be recorded at 2 minutes, 5 minutes and thereafter at 10 minutes interval throughout the course of surgery.

DRUGS

All drugs that will be used in this study will be those licensed for clinical use in Nigeria and they include:

0.25% plain bupivacaine, dexamethasone, chlorpheniramine, atropine, paracetamol and diclofenac. All drugs will be provided by the researcher.

PERIOD OF STUDY This study will be done over a period of about 3-6 months DATA MANAGEMENT Based on the calculation of sampled size, 96 patients would be In 2 groups of 48 patients each.

Data collection will be done with a proforma in section A-D

DATA ANALYSIS Data will be analysed using statistic package for social science (SPSS) version 15 Demographic variable will be represented with tables and charts while summary statistics will be done with means and proportions.

Test of association for categorical variables will be done using chi square. Test of association for quantities will be done using t tests and anova. Level of statistical significance will be set at p value of < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-6 years, classified as American Society of Anesthesiologist (ASA) 1 and 11 who are undergoing herniotomy and whose parents or legal guardian has duly signed an informed consent form.

Exclusion Criteria:

* Patients with hypersensitivity to any local anesthetics
* Children with Bleeding diathesis
* Presence of Infections at puncture sites
* Preexisting neurological disease
* Patients with diabetes mellitus
* Failure to consent by parents

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
time to first analgesic requirement | within the first 24 hours post operatively
  defined as the time from the caudal injection till the first rescue analgesia was administered (Modified Objective Pain Score, mOPS score of 4 or more).

SECONDARY OUTCOMES:
the number of oral paracetamol | required in the first 24 hours post operatively

OTHER OUTCOMES:
Postoperative pain will be assessed using a modified Objective Pain Score (mOPS) every 30 min for the first 2 h and at 4, 6, 8, 10, 12, 18, and 24 h postoperatively | within 24 hours
Motor block will be assessed using a modified Bromage scale consisting of four points [0 = full motor strength (flexion of knees and feet), 1 = flexion of knees, 2 = little movement of feet only, 3 = no movement of knees or feet | within 24 hours
The sedation score will; be assessed using a four-point scale (1, alert and aware; 2, asleep, arousable by verbal contact; 3, asleep, arousable by physical contact; and 4, asleep, not arousable). | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: FAGBOHUN A OMOLOLA, MBBS, Principal Investigator — SCHOOL OF ANAESTHETIC STUDIES BADAGRY